CLINICAL TRIAL: NCT04714606
Title: Feasibility Controlled Trial of an 8-session Group Intervention for Siblings of Children Who Have ASD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Surrey (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 260159
Record Dates: First submitted 2020-12-09; First posted 2021-01-19 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sibling support group (Experimental): 8 session, tailored support group for siblings of children who have an ASD
  Interventions: Other: Sibling support group
- Booklet (Active Comparator): Control condition in which siblings of children who have an ASD will receive a tailored booklet to complete at home
  Interventions: Other: None - control condition

INTERVENTIONS:
Other: Sibling support group — The intervention is a novel, 8 session sibling support group which has been created for the purpose of the study.
  Arms: Sibling support group
Other: None - control condition — The second arm of the study is a control condition in which participants will be given a tailored booklet to complete at home as it was deemed unethical to provide them with nothing.
  Arms: Booklet

SUMMARY:
A feasibility controlled trial of an eight-session group intervention for siblings of children who have an Autism Spectrum Disorder (ASD).

Children will be recruited from a multi-academy trust of nine schools. Due to the on-going impact of COVID-19 restrictions, children will be allocated to the intervention condition (eight session support group) if they are physically attending school and to the control condition (receipt of a booklet) if they remain at home. Pre and post outcome measures will be completed by children and their parents in both research arms.

ELIGIBILITY:
Inclusion Criteria:

1. 7-11 years old.
2. Must have a sibling who has a formal diagnosis of ASD.
3. Must be competent in the English language.
4. Must be in mainstream education.
5. Must be willing and able to engage in an eight-session group intervention (including being accompanied to and from the group by their parents/carers).
6. Must be registered with a GP and parental consent gained to inform the GP that the sibling is attending the group.

Exclusion Criteria:

1. If the sibling has a diagnosis of ASD themselves.
2. If there are any clear risk concerns (e.g. any thought or intent to harm self or others, involvement in court proceedings or with the criminal justice system).
3. If the sibling is currently receiving any other psychological treatment.
4. If the sibling has a learning disability or difficulty that will make it hard to access the group content and/or capacity to provide informed consent.

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Change in Strengths & Difficulties Questionnaire (SDQ, Goodman et al., 2009) scores | Pre (Week 1) and post (Week 6) intervention
  Questionnaire used to measure effectiveness pre and post intervention or control condition. Lower scores indicate better outcome.
Change in Paediatric Quality of Life Inventory (PedsQL V4.0; Varni, Seid & Kurtin, 2001) scores | Pre (Week 1) and post (Week 6) intervention
  Questionnaire used to measure effectiveness pre and post intervention or control condition. Higher scores indicate better outcome.
Change in Knowledge of Autism Questionnaire (KAS; Ross & Cuskelly, 2006) scores | Pre (Week 1) and post (Week 6) intervention
  Questionnaire used to measure knowledge of autism pre and post intervention or control condition. Higher scores indicate better outcome.
Change in Goal Based Outcomes (GBOs, Law & Jacob, 2015) scores Goal Based Outcomes (GBOs, Law & Jacob, 2015) | Pre (Week 1) and post (Week 6) intervention
  Questionnaire used to measure effectiveness pre and post intervention or control condition. Higher scores indicate better outcome.

SECONDARY OUTCOMES:
Experience of Service Questionnaire (ESQ, Attride-Stirling, 2002) | Post intervention (6 weeks after Time 1)
  Questionnaire used to measure experience post intervention or control condition. Higher scores indicate better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Lucy Ms Watson, Principal Investigator — University of Surrey
Locations (1):
- The Howard Partnership Multi-Academy Trust, Leatherhead, United Kingdom

IPD SHARING:
Plan to Share IPD: No